CLINICAL TRIAL: NCT06078670
Title: Phase Ib/II Clinical Study of PARP Inhibitor CVL218 in Combination With Therapy in Patients With Advanced Solid Tumors
Brief Title: PARP Inhibitor CVL218 in Combination Therapy for Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL218-1003
Record Dates: First submitted 2023-09-18; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor
Keywords: Triple negative breast cancer; stomach cancer; Intestinal cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Stomach Neoplasms; Intestinal Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Triple Negative Breast Cancer (Experimental): CVL218+Toripalimab+Paclitaxel For Injection (Albumin Bound)
  Interventions: Drug: CVL218
- Stomach cancer (Experimental): CVL218+Sintilimab+Paclitaxel Injection
  Interventions: Drug: CVL218
- Intestinal cancer (Experimental): CVL218+Sintilimab+Fruquintinib
  Interventions: Drug: CVL218

INTERVENTIONS:
Drug: CVL218 — Arm1: Triple negative breast cancer CVL218 is administered orally Triplelizumab injection was administered intravenously (IV) 240mg on D1 Paclitaxel injection (Kealil) 125mg /m2, D1, D8 administration Every 21 days for a drug cycle; Arm2: Gastric cancer CVL218 is administered orally Sindilizumab injection was given intravenously (IV) 200mg on D1 Paclitaxel injection (Taxol) 175mg /m2, D1 administration Every 21 days for a drug cycle; Arm3: Intestinal cancer CVL218 is administered orally Sindilizumab injection was given intravenously (IV) 200mg on D1 Fuquinitinib capsule 5mg QD orally, D1-14 administration Every 21 days is a medication cycle.
  Other Names: Toripalimab、Paclitaxel For Injection (Albumin Bound)、Sintilimab、Paclitaxel Injection、Fruquintinib

SUMMARY:
This study aims to evaluate the efficacy of CVL218 in combination with Toripalimab injection/Sintilimab injection (Darbersol, Sintilimab) in the treatment of advanced solid tumors. It focuses on assessing the safety, tolerability, and pharmacokinetic profile of a three-drug combination regimen comprising albumin-bound paclitaxel injection (Kealil), paclitaxel injection (Taxol), and Fuquinitinib capsule (Aiutec, Fruquintinib).

DETAILED DESCRIPTION:
This Phase Ib/II clinical study is designed to determine the recommended Phase II dosage of the combination therapy and its initial efficacy. The study consists of two phases: an exploratory phase (Ib) and an extended phase (II), each divided into three stages: the screening period, treatment period, and follow-up period.

The screening period occurs 28 days prior to the first dose administration. Three parallel queues were organized, with Phase Ib enrolling 3-6 participants per dose level cohort and Phase II enrolling approximately 20 participants per cohort.

In Phase II, subjects must demonstrate evidence of deleterious HRD gene variants (such as BRCA1, BRCA2, PALB2, ATM, CHEK2 variants) or a positive PD-L1 molecular expression level combined score (CPS) of ≥1. Additionally, Phase II participants are required to consent to the provision of sufficient archived or fresh tumor tissue and blood samples for biomarker analysis in the central laboratory, including determination of HRD gene mutation status and PD-L1 expression level (details in Section 7.4).

During the treatment period, the three cohorts received CVL218 orally (PO) in combination with a fixed dose of either terriplizumab injection (Toripalimab) or Sintilimab injection (Darbersol, Sintilimab). Additionally, they were administered albumin-bound paclitaxel injection (Kealil)/paclitaxel injection (Taxol)/Fuquintinib capsule (Aiutec, Fruquintinib).

CVL218 was administered at two dose levels, ranging from low to high (500 mg, 700 mg), twice daily (BID), during the exploration of cohorts in Phase Ib. After determining the recommended dose of CVL218 in all cohorts of the three-drug combination, this dose level was maintained during Phase II. When CVL218 and the combination were administered on the same day, CVL218 was given first.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients between the ages of 18 and 75 (including those aged 18 and 75, and those over 60 years old should not suffer from more than 3 complications of heart, lung, liver and kidney function at the same time), regardless of gender.

  2. Patients with locally advanced or metastatic advanced solid tumors confirmed by histology or cytology (including but not limited to triple-negative breast cancer, gastric cancer, colorectal cancer); Patients with ≤1 line of standard treatment failure (disease progression after treatment or intolerability of toxic side effects of treatment), or no standard treatment, or unable to receive standard treatment.

  3. In stage II, patients with positive PD-L1 molecular expression level combined with CPS≥1 were required to be enrolled, or there was evidence of harmful HRD gene variants (BRCA1, BRCA2, PALB2, ATM, CHEK2 variants, etc.).

Exclusion Criteria:

* Chemotherapy, radiotherapy, biotherapy and endocrinology were received within 4 weeks before the first administration

Treatment, immunotherapy and other antitumor drugs, except the following:

Nitrosourea or mitomycin C within 6 weeks before first use of the study drug;

Oral fluorouracil and small molecule targeted drugs are used before first investigational drugs

2 weeks or within 5 half-lives of the drug, whichever is longer;

Traditional Chinese medicines with anti-tumor indications were used within 2 weeks before the first use of study drugs.

2. Received other investigational drugs or treatments that are not on the market within 4 weeks prior to initial administration

Therapy.

3. Received major organ surgery (excluding puncture) within 4 weeks prior to initial administration

Biopsy) or significant trauma.

4. Received systemic glucocorticoids (strong) within 14 days prior to initial administration

Pine > 10mg/ day or equivalent dose of similar drugs) or other immunosuppressant

Treatment;

Except in the following cases: topical, ocular, intraarticular, intranasal, and inhalation

Type I glucocorticoid therapy; Short-term use of corticosteroids for prophylactic treatment (eg to prevent contrast allergy).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) during the observation period of DLT | Incidence of dose-limiting toxicity (DLT) during the observation period of DLT，No more than six months；The interruption and reduction of drug dose in the cohorts of the combination regimen were studied，No more than three years
  The duration of DLT evaluation in Phase Ib is within the first cycle after dosing (within 21 days). Starting from the 500mg BID CVL218 dose group, each dose group was enrolled on the basis of 3 cases. If DLT was present in 2/3 or more of the group, one dose level should be lowered. If 1/3 of the subjects developed DLT, 3 more subjects were enrolled with the same dose. If 2/6 or more subjects develop DLT, the dose level should be lowered by one dose. After each dose group completes the DLT assessment, it is decided whether to move to the next dose group. The recommended dose (RP2D) will be determined based on the combined data of safety and tolerability, PK, pharmacodynamics, and initial anti-tumor efficacy of the drug obtained during the dose escalation phase. If dose-limiting toxicity (DLT) occurs in 0/3 subjects in a group, or in less than 2/6 subjects, the CVL218 dose can be used as the recommended dose.

SECONDARY OUTCOMES:
Duration of response (DoR), progression-free survival (PFS), disease control rate (DCR)as assessed by the RECIST v1.1 | Imaging evaluation was performed every 6 weeks (±7 days) for six months prior to treatment. After six months, they were evaluated every 12 weeks (±7 days). Tumor evaluation can be performed more frequently by the investigator according to clinical needs.
  Duration of response (DoR), progression-free survival (PFS), disease control rate (DCR)as assessed by the RECIST v1.1

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.